CLINICAL TRIAL: NCT00617526
Title: A Multicenter Phase 2a, Randomized, Double-blind, Placebo-controlled, Proof-of-concept Trial to Determine the Antiviral Activity, Pharmacokinetics, Tolerability and Safety of RDEA806 in HIV-1 Positive, Antiretroviral naïve Subjects
Brief Title: Naïve HIV POC Monotherapy Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ardea Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RDEA806-201
Record Dates: First submitted 2008-02-06; First posted 2008-02-18 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2013-12

CONDITIONS: HIV Infections
Keywords: HIV; treatment naïve
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- RDEA806 400 mg (Experimental): Placebo or RDEA806 400 mg twice daily (BID) for 7 days and a single morning dose on Day 8.
  Interventions: Drug: RDEA806 400 mg; Drug: Placebo
- RDEA806 600 mg (Experimental): Placebo or RDEA806 600 mg once daily (QD) for 7 days with an additional dose on the morning of Day 8.
  Interventions: Drug: Placebo; Drug: RDEA806 600 mg
- RDEA806 800 mg (Experimental): Placebo or RDEA806 800 mg QD using enteric coated tablets for 7 days with an additional morning dose on Day 8.
  Interventions: Drug: Placebo; Drug: RDEA806 800 mg
- RDEA806 1000 mg (Experimental): Placebo or RDEA806 1000 mg QD using enteric coated tablets for 7 days with an additional dose on the morning of Day 8.
  Interventions: Drug: Placebo; Drug: RDEA806 1000 mg

INTERVENTIONS:
Drug: RDEA806 400 mg
  Arms: RDEA806 400 mg
Drug: Placebo — Placebo
Drug: RDEA806 1000 mg
  Arms: RDEA806 1000 mg
Drug: RDEA806 600 mg
  Arms: RDEA806 600 mg
Drug: RDEA806 800 mg
  Arms: RDEA806 800 mg

SUMMARY:
The primary objective of the trial is:

• to evaluate the change from baseline in plasma viral load with placebo and one of up to 4 dose regimens of RDEA806.

The secondary objectives are:

Efficacy

* to describe the nadir of the plasma viral load
* to describe the DAVG
* to assess the proportion of subjects who reached a drop in viral load of 0.5 log, 1 log, or reach an undetectable viral load
* to assess the plasma viral load decay rate
* to evaluate immunologic changes (as measured by CD4 and CD8 cells)
* to evaluate the genotypic and phenotypic pattern of the virus Pharmacokinetics
* to evaluate the pharmacokinetics and the pharmacokinetic/pharmacodynamic relationship of RDEA806 Safety
* to evaluate the safety and tolerability of bid and qd dosing of RDEA806 as monotherapy

ELIGIBILITY:
Inclusion Criteria:

* Documented chronic HIV-1 infection
* HIV-1 plasma viral load at screening visit above 5000 HIV-1 RNA copies/ml
* Male, aged above 18 years and less than 65 years of age
* Adequate method of birth control
* Subject has never received an antiretroviral agent (NRTI, NNRTI, PI, entry inhibitor or integrase inhibitor) for the treatment of HIV and agrees not to start antiretroviral therapy prior to enrollment or subject has only received a short course of treatment for less than 14 days and has been off treatment for at least 8 weeks
* Subject has no primary mutation in the reverse transcriptase (RT) gene associated with resistance to RT inhibitors and no major mutation in the protease gene associated with resistance to PIs determined by genotypic resistance testing at screening

Exclusion Criteria:

* History or suspicion of alcohol or drug abuse which in the Investigator's opinion may lead to non-compliance
* CD4 count < 350 cells/mm3
* Life expectancy of less than 6 months
* Receipt of an investigational drug within 30 days prior to the trial drug administration
* Receipt of any vaccine within 30 days of screening visit
* Acute HIV-1 infection (seroconversion illness)
* Acute hepatitis A or acute or chronic hepatitis B or C infection
* Currently active acquired immune deficiency syndrome (AIDS)-defining illness (Category C conditions according to the Centers for Disease Control [CDC] Classification System for HIV Infection 1993)
* No clinically relevant laboratory abnormalities Renal impairment: serum creatinine > 1.5 x ULN
* Febrile illness within 120 hours prior to dosing
* History of severe drug allergy or hypersensitivity
* Significant cardiac dysfunction

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2008-01; Primary Completion 2008-06 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HIV plasma viral load | 9 days

SECONDARY OUTCOMES:
Safety will be assessed as adverse and HIV related events, clinical laboratory test results(hematology, chemistry, urinalysis), vital signs, 12-lead electrocardiograms (ECGs), and physical examination | 22 days
Pharmacokinetics and Resistance | 22 days

CONTACTS AND LOCATIONS:
Overall Officials: Vijay Hingorani, MD, PhD, Study Director — Ardea Biosciences
Locations (2):
- Hamburg, Germany
- London, United Kingdom

REFERENCES:
- [Derived] Moyle G, Boffito M, Stoehr A, Rieger A, Shen Z, Manhard K, Sheedy B, Hingorani V, Raney A, Nguyen M, Nguyen T, Ong V, Yeh LT, Quart B. Phase 2a randomized controlled trial of short-term activity, safety, and pharmacokinetics of a novel nonnucleoside reverse transcriptase inhibitor, RDEA806, in HIV-1-positive, antiretroviral-naive subjects. Antimicrob Agents Chemother. 2010 Aug;54(8):3170-8. doi: 10.1128/AAC.00268-10. Epub 2010 May 24. PMID 20498326